CLINICAL TRIAL: NCT00724763
Title: The Effect of Acupuncture on Blood Pressure and HRV
Brief Title: The Effect of Acupuncture on Blood Pressure and Heart Rate Variability (HRV)
Acronym: Acupuncture
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: John Zhang, MD, PhD, Logan University, College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD0609080136
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Hypertension
Keywords: acupuncture, high blood pressure, HRV
MeSH Terms: conditions — Hypertension | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatment group.
  Interventions: Device: acupuncture
- 2 (Sham Comparator): control group
  Interventions: Device: sham needle treatment

INTERVENTIONS:
Device: acupuncture — to Liv 3 and PE 9.
  Arms: 1
Device: sham needle treatment — needle not in meridian area
  Arms: 2

SUMMARY:
This research is designed to study the effects of needle acupuncture on blood pressure and HRV by stimulating certain acupuncture points and meridians.

DETAILED DESCRIPTION:
Outcome measurements include blood pressure and heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Male or female suffering from mild hypertension (systolic BP between 130-165 mmHg, diastolic BP between 90-120 mmHg).

Exclusion Criteria:

* Individuals with heart, kidney, thyroid disorders, diabetes, chronic disease or illness, neurological diseases, skin or bleeding disorders,
* Currently taking prescription or OTC medications and/or herb/supplements that effect BP or autonomic tone will not be recruited into the study.
* In addition, individuals who have a pacemaker and/or are pregnant will not be recruited in the study. A health history questionnaire was used to screen subjects.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Blood pressure and HRV | five weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Logan University, Chesterfield, Missouri, United States